CLINICAL TRIAL: NCT00866801
Title: Cardiac Sympathetic Innervation and Coronary Blood Flow Regulation During General Anesthesia
Brief Title: Coronary Blood Flow Regulation During General Anesthesia
Status: Completed | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Netherlands Heart Foundation (Other)
Responsible Party: Principal Investigator, C.S.E. Bulte, MD, Amsterdam UMC, location VUmc
Other Study IDs: ANES 2008-12; 2008 T003
Record Dates: First submitted 2009-03-20; First posted 2009-03-23 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Myocardial Ischemia; Autonomic Neuropathy; Healthy; Diabetes
Keywords: coronary blood flow; coronary flow reserve; cardiac sympathetic innervation; general anesthesia; thoracic epidural; autonomic dysfunction; autonomic neuropathy
MeSH Terms: conditions — Myocardial Ischemia; Diabetes Mellitus; Primary Dysautonomias

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Frozen plasma will be retained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Healthy: Healthy subjects scheduled for general anesthesia
- Healthy with thoracic epidural anelgesia: Healthy subjects scheduled for general anesthesia and thoracic epidural analgesia
- Diabetes: Subjects with diabetes scheduled for general anesthesia
- Diabetes with autonomic neuropathy: Subjects with diabetes and cardiovascular autonomic neuropathy scheduled for general anesthesia

SUMMARY:
The central hypothesis in the present project is that general anesthesia may alter autonomic control such that perioperative coronary blood flow (CBF) is significantly disturbed.

These disturbances in coronary blood flow may contribute to the development of myocardial ischemia in the perioperative period. Furthermore, patients with an intrinsically altered autonomic sympathetic innervation, like diabetics, are even more prone to develop perioperative disturbances in coronary blood flow.

Here the researchers will investigate what the direct effects are of general and locoregional anesthesia on the CBF. Furthermore, the researchers aim to evaluate whether diabetic subjects show more disturbed CBF responses to anesthesia as compared to non-diabetics.

DETAILED DESCRIPTION:
In response to intraoperative stress, increased autonomic sympathetic activity may alter myocardial oxygen demand. Under normal physiological circumstances, sympathetic stimulation increases myocardial blood flow via adrenergic coronary vasodilation. However, coronary vessels contain both α- and β-adrenoreceptors, and if the coronary circulation is impaired due to cardiovascular disease, unopposed adrenergic coronary vasoconstriction may contribute to ischemia. Anesthetics reduce both coronary blood flow (CBF) regulation and the sympathetic autonomic nervous activity. However, it is unclear whether anesthetic-related reductions in CBF are a result of inhibited autonomic sympathetic innervation. Data regarding alterations in myocardial blood flow in response to sympathetic stimulation during anesthesia provide conflicting results. Moffitt and Sethna showed in patients undergoing cardiac surgery that CBF decreased during sternotomy-induced sympathetic stimulation, whereas Kirno et al. showed an increase in coronary blood flow after sternotomy. To our best knowledge, coronary vascular responses to sympathetic stimulation in anesthetized healthy humans are lacking because of absence of reliable non-invasive measurement of myocardial blood flow. The introduction of non-invasive contrast-echocardiographic techniques that allow evaluation of regional myocardial blood flow enable evaluation of the relation between autonomic control and CBF during anesthesia.

Cardiac complications like myocardial ischemia remain one of the main causes of perioperative morbidity and mortality. Interestingly, the presence of cardiovascular autonomic neuropathy (CAN) strongly predicts abnormalities in myocardial perfusion and impaired coronary vasodilator responses to stress. This implies that symptoms of CAN, like resting tachycardia, orthostasis and alterations in heart rate variability may predict the degree of impairment of CBF regulation. Indeed, autonomic neuropathy as determined by heart rate variability predicted mortality in patients with coronary artery disease undergoing non-cardiac surgery, but the contribution of impaired coronary vasodilatory responses to these results has not been established. Clarification of the relation between autonomic control and CBF during anesthesia may not only contribute to our insight in pro-ischemic processes in the heart, but may lead to changes in preoperative assessment of patients at risk for perioperative ischemia, thereby reducing perioperative complications.

ELIGIBILITY:
Inclusion Criteria:

* male
* age between 18-75 years
* scheduled for non-cardiac intermediate or high risk surgery
* for patient group 2: indication for thoracic epidural anesthesia

Exclusion Criteria:

* neurosurgery
* known/documented cardiac disease
* (untreated) hypertension
* abnormal ECG or echocardiogram
* peripheral vascular disease
* renal disease requiring hemo- or peritoneal dialysis
* inability to perform transthoracic echocardiography
* medication interfering with presynaptic catecholamine uptake
* for patient group 2: contra-indication for thoracic epidural anesthesia (bleeding diathesis, infection at the puncture site, patient refusal, severe stenotic valvular disease)
* previous allergic reaction to echocardiographic contrast agents
* contraindications for the use of echocardiographic contrast agents

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists patients scheduled for surgery and general anesthesia. Patients will be recruited from the preoperative screening clinic in the four, aforementioned, groups of patients.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2009-04; Primary Completion 2014-02 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Coronary flow reserve | Within the first 3 days postoperatively

SECONDARY OUTCOMES:
Diabetic autonomic neuropathy | Within the first 3 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Carolien SE Bulte, MD, Principal Investigator — Amsterdam UMC, location VUmc; R. A. Bouwman, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc; C. Boer, PhD, Study Chair — Amsterdam UMC, location VUmc; S. A. Loer, MD, PhD, MSC, Study Director — Amsterdam UMC, location VUmc; O. Kamp, MD, PhD, Study Chair — Amsterdam UMC, location VUmc; M. Diamant, MD, PhD, Study Chair — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] Bulte CS, van den Brom CE, Loer SA, Boer C, Bouwman RA. Myocardial blood flow under general anaesthesia with sevoflurane in type 2 diabetic patients: a pilot study. Cardiovasc Diabetol. 2014 Mar 23;13:62. doi: 10.1186/1475-2840-13-62. PMID 24656118